CLINICAL TRIAL: NCT01407848
Title: Trial on Treatment With Inhaled Furosemide of Preterm and Term Neonates With Transient Tachypnoea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Patrizia Nitsch-Felsecker, Dr. med., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-1488; 2011-003473-29 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-08-02 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Transient Tachypnoea of the Newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furosemide (Experimental): 1 mg/kg/Ed
  Interventions: Drug: Furosemide
- Saline 0,9% (Active Comparator): 1ml/kg/Ed
  Interventions: Drug: Saline 0,9%

INTERVENTIONS:
Drug: Furosemide — Patients received nebulised Furosemide iv solution 1 mg/kg (4x/d) for max.3 consecutive days.
  Other Names: inhaled furosemide
  Arms: Furosemide
Drug: Saline 0,9% — nebulised 0,9% saline 4x/d for max.3 days
  Other Names: natrium chloride
  Arms: Saline 0,9%

SUMMARY:
In this study we will prospectively analyze the benefit of inhaled furosemide for preterm and term neonates with Transient Tachypnoea.

DETAILED DESCRIPTION:
In this study we will prospectively analyze the benefit of inhaled furosemide for preterm and term neonates with transient Tachypnoea. Patients received nebulised Furosemide iv solution 1 mg/kg or nebulised 0,9% saline (4x/d) under blind conditions in random order so long as need a CPAP-treatment but max. 3 days. 20 Patient will be treating.

The benefit will be measured as reduction of dyspnea, respiratory rate, oxygen demand and time on CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with 35+0-39+0 GA on the first day of life with the clinical diagnosis of Transient Tachypnoea
* The need for CPAP >6 h to obtain the oxygen saturation >92%
* Written informed consent of parent/guardian

Exclusion Criteria:

* Systemic infection
* Intubation and mechanical ventilation before Inclusion in the trail
* Malformation and any other several disease with disturb of respiratory
* Subjects participating in other clinical trials

Min Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reduction of the Silverman-Score | 0-72 h or up to end of CPAP after start of the study
  The primary endpoint of the study is the reduction of the Silverman score as an indicator of respiratory distress of the infant.
  Silverman Score is the standard score to describe the degree of respiratory distress of neonate.

SECONDARY OUTCOMES:
Oxygen supplementation | 0-72 h or up to end of CPAP after start of the study
A need for secondary intubation and mechanical ventilation | 1-3 day of life
body weight | 1-3 day of life
CPAP-time | 0-72 h or up to end of CPAP after start of the study
blood electrolytes (Na+, K+, Ca++, HCO3-, Cl-) | 0-72 h after start of the study
blood gas (pH, pCO2,pO2) | 0-72 h after start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Roth, Prof. Dr., Principal Investigator — University Cologne
Locations (1):
- Children´s Hospital University of Cologne, Cologne, North Rhine-Westphalia, Germany